CLINICAL TRIAL: NCT02499497
Title: A Selective Androgen Receptor Modulator for Symptom Management in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Shalender Bhasin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-120
Record Dates: First submitted 2015-07-06; First posted 2015-07-16 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LY2452473

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Subjects who meet the eligibility criteria, will be randomized, to either placebo, LY SARM Dose 1, LY SARM Dose 2 or LY SARM Dose 3 daily, oral per cycle.
  Interventions: Drug: Placebo
- LY2452473 Dose 1 (Active Comparator): Subjects who meet the eligibility criteria, will be randomized, to either placebo, LY SARM Dose 1, LY SARM Dose 2 or LY SARM Dose 3 daily, oral per cycle.
  Interventions: Drug: LY2452473
- LY2452473 Dose 2 (Active Comparator): Subjects who meet the eligibility criteria, will be randomized, to either placebo, LY SARM Dose 1 or LY SARM Dose 2 or LY SARM Dose 3 daily, oral per cycle.
  Interventions: Drug: LY2452473
- LY2452473 Dose 3 (Active Comparator): Subjects who meet the eligibility criteria, will be randomized, to either placebo, LY SARM Dose 1, LY SARM Dose 2 or LY SARM Dose 3 daily, oral per cycle.
  Interventions: Drug: LY2452473

INTERVENTIONS:
Drug: LY2452473 — LY2452473 is a selective androgen receptor modulator which is agonist on the muscle but which spares the prostate.
  Other Names: Selective Androgen Receptor Modulator
  Arms: LY2452473 Dose 1; LY2452473 Dose 2; LY2452473 Dose 3
Drug: Placebo — The participants will receive pills containing no active drug.
  Other Names: Inactive comparator
  Arms: Placebo

SUMMARY:
This research study is studying the use of a targeted therapy called LY SARM, which is an investigational drug from a new class of molecules called Selective Androgen Receptor Modulators (SARMs) as a possible improvement in quality of life for participants who have undergone radical prostatectomy. Androgens are a group of hormones that play a role in male traits and reproductive activity.

The names of the study interventions involved in this study are:

- LY2452473

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved LY SARM/LY2452473 as a treatment for any disease.

In this research study, the investigators are studying a new investigational drug called LY SARM (LY2452473). Concerns about the potential adverse effects of testosterone on the prostate have led to the development of molecules called SARMs (Selective Androgen Receptor Modulators). This investigational drug may improve sexual function, quality of life, muscle and bone mass in men with prostate cancer. This molecule was chosen because there is some evidence that shows it may help to improve sexual function and aid in the improvement of muscle mass while not having any influence on the prostate.

ELIGIBILITY:
Inclusion Criteria

* Age 19 years of age or older
* History of prostate cancer

  * Stage pathological tumor-2 (pT2) N0, M0 lesions (If American Joint Committee on Cancer (AJCC) staging is not available in medical records, the investigators will infer the staging based on extensive review of the pathology report)
  * Combined Gleason score < 7 (3+4)
  * Radical prostatectomy two or more years ago
  * Preoperative prostate-specific antigen (PSA)<10 ng/ml (if pre-operative PSA is not available in medical records, low-risk subjects with a Gleason score of 6(3+3) and who are at least 5 years out of surgery will be considered for enrollment)
  * PSA <0.1 ng/mL using an assay that has a functional sensitivity of 0.1 ng/mL for at least two years after radical prostatectomy
* Serum testosterone, measured by Liquid chromatography-tandem mass spectrometry (LC-MS/MS), <300 mg/dL and/or free testosterone by equilibrium dialysis <60 pg/mL.

  * Derogatis Index of Sexual Function Male II (DISF-M-II) score ≤20, fatigue (FACIT-F score <30), or physical dysfunction (self-reported difficulty in walking a 1/4 mile or climbing two flights of stairs, short physical performance battery score 4 to 9).
* Ability to understand and the willingness to sign a written informed consent document.

  * Agree to use adequate contraception prior to receiving the study drug, for the duration of study participation, and 4 months after completion of LY SARM administration.

Exclusion Criteria

* History of radiation monotherapy
* History of androgen deprivation therapy
* Use of testosterone, dehydroepiandrosterone (DHEA), estrogens, gonadotropin-releasing hormone (GnRH) analogs, antiandrogens, spironolactone, ketoconazole, recombinant human growth hormone (rhGH), or megestrol acetate within the past 6 months
* Use of prednisone 20 mg daily or equivalent doses of other glucocorticoids for more than two weeks within the past 6 months
* Use of Clarithromycin, telithromycin, chloramphenicol, itraconazole, nefazodone, cobicistat within the past 6 months
* Use of penile implants, vacuum pump devices, intra-cavernosal injections
* Hematocrit >50%
* Serum creatinine >2.5 mg/dL
* Aspartate aminotransferase (AST) greater than 3x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) greater than 3x ULN
* Hemoglobin A1c >7.5%
* Body mass index (BMI) >40 kg/m2
* Diabetes requiring insulin therapy
* Severe untreated sleep apnea (treatment is defined as therapy with continuous positive airway pressure (CPAP), BiPAP, adaptive servo-ventilation (ASV), or other positive air pressure device)
* Uncontrolled heart failure (NYHA class 3 or 4)
* History of HIV
* Myocardial infarction within the last 3 months
* Acute coronary syndrome within the last 3 months
* Revascularization surgery within the last 3 months
* Stroke within the last 3 months
* Diagnosed schizophrenia or bipolar disorder or untreated depression
* Not appropriate for study based on physician discretion

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - John Hopkins Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center (Referring site only), Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Pencina KM, Burnett AL, Storer TW, Guo W, Li Z, Kibel AS, Huang G, Blouin M, Berry DL, Basaria S, Bhasin S. A Selective Androgen Receptor Modulator (OPK-88004) in Prostate Cancer Survivors: A Randomized Trial. J Clin Endocrinol Metab. 2021 Jul 13;106(8):2171-2186. doi: 10.1210/clinem/dgab361. PMID 34019661

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: The participants will receive pills containing no active drug daily for 12-weeks.
- LY2452473 Dose 1: The participants will receive 1 mg LY2452473 daily for 12-weeks.
  N-[(2S)-7-cyano-1,2,3,4-tetrahydro-4-(2-pyridinylmethyl)cyclopent[b]indol-2-yl]-,1-methylester (LY2452473): LY2452473 is a selective androgen receptor modulator which is agonist on the muscle but which spares the prostate.
- LY2452473 Dose 2: The participants will receive 5 mg LY2452473 daily for 12-weeks.
  LY2452473: LY2452473 is a selective androgen receptor modulator which is agonist on the muscle but which spares the prostate.
- LY2452473 Dose 3: The participants will receive 15 mg LY2452473 daily for 12-weeks.
  LY2452473: LY2452473 is a selective androgen receptor modulator which is agonist on the muscle but which spares the prostate.
Period: Overall Study
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Started | 36 | 28 | 36 | 14
Completed | 32 | 22 | 35 | 13
Not Completed | 4 | 6 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- LY2452473 Dose 1: The participants will receive 1 mg LY2452473 daily for 12-weeks.
  LY2452473: LY2452473 is a selective androgen receptor modulator which is agonist on the muscle but which spares the prostate.
- Total: Total of all reporting groups
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3 | Total
Number analyzed (Participants) | 36 | 28 | 36 | 14 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (6.1) | 67.1 (7.87) | 67.4 (8.6) | 69.6 (7.1) | 67.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 36 | 28 | 36 | 14 | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 28 | 36 | 14 | 114
Weight [Mean (Standard Deviation); unit: kg] | 84.9 (12.7) | 92.7 (10.7) | 89.7 (15.4) | 86.7 (12.5) | 88.5 (13.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (3.8) | 29.8 (3.89) | 29.3 (4.1) | 29.2 (5.1) | 29.0 (4.1)
Short Physical Performance Battery (SPPB) score [Mean (Standard Deviation); unit: units on a scale] — The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. The scores range from 0 to 12. The higher the score, the better the performance.
  units on a scale | 11.4 (1.15) | 11.1 (1.21) | 11.1 (1.42) | 11.1 (1.07) | 11.2 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sexual Activity Score of Psychosexual Daily Questionnaire (PDQ-4)
Description: The primary outcome is change in sexual activity score, assessed by the Psychosexual Daily Questionnaire (PDQ). The questionnaire covered 3 different domains: 1) sexual desire, enjoyment, and performance; 2) sexual activity score; and 3) mood. Sexual activity was assessed using a checklist format (12-item) and the score range of 0 to 12 with higher scores representing better sexual activity.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 28 | 23 | 35 | 13
units on a scale | 0.04 (0.19) | 0.45 (0.26) | -0.02 (0.22) | 0.12 (0.27)

2. Secondary Outcome: Change in All Domains of International Index of Erectile Function (IIEF)
Description: IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 12
units on a scale
  Erectile Function | 2.34 (1.02) | 0.92 (0.48) | -0.50 (0.94) | 3.38 (2.83)
  Intercourse satisfaction | 0.97 (0.50) | 0.42 (0.25) | -0.22 (0.39) | 0.92 (1.59)
  Orgasmic function | 0.12 (0.48) | 0.17 (0.32) | -0.53 (0.57) | 0.75 (0.85)
  Sexual desire | 0.30 (0.22) | 0.46 (0.38) | -0.19 (0.25) | 0.83 (0.61)
  Overall satisfaction | 1.13 (0.34) | 0.79 (0.32) | 0.31 (0.33) | 0.25 (0.70)
  Composite IIEF | 4.79 (1.96) | 2.73 (1.28) | -1.22 (1.90) | 6.14 (5.90)

3. Secondary Outcome: Change in Sexual Activity, Interest, and Desire Scale (SAID)
Description: The Sexual Activity, Interest, and Desire Scale (SAID) is an 8-item questionnaire that evaluates 3 response domains, including sexual thinking, sexual arousal, and sexual activity. The score was linearly transformed to a 0 to 100 scale for each item. The average score ranges 0-100. The higher the score, the better the sexual function.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 12
units on a scale | -0.67 (2.36) | 4.25 (2.85) | -3.00 (3.27) | -1.50 (4.67)

4. Secondary Outcome: Change in Derogatis Index of Sexual Function Male II (DISF-M-II)
Description: Derogatis Index of Sexual Function Male II (DISF-M-II) is a 25-item questionnaire that provides an estimate of perceived quality of sexual activities in 5 response domains: sexual desire/drive (range 0-33), sexual arousal (range 0-33), sexual activity (range 0-35), orgasm (range 0-26), and sexual satisfaction/partner relationship (range 0-25). The total possible score (sum of 5 domains) range of 0 to 152 with higher scores representing better function.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 23 | 36 | 12
units on a scale
  Sexual Desire | -0.88 (0.89) | 0.87 (1.63) | -0.81 (0.97) | 1.08 (2.21)
  Sexual Arousal | 0.45 (0.62) | 0.83 (0.74) | 0.00 (0.74) | 0.67 (0.94)
  Sexual Activity | -0.33 (0.65) | 0.96 (0.81) | 0.53 (0.67) | 0.67 (0.83)
  Orgasm | 0.55 (0.82) | 0.57 (0.84) | -0.31 (0.77) | 0.75 (2.07)
  Sexual Satisfaction | 0.27 (0.69) | 1.22 (1.18) | 0.22 (0.91) | 1.42 (1.69)
  Composite DISF-M-II | 0.06 (2.70) | 4.43 (3.91) | -0.36 (3.26) | 4.58 (5.98)

5. Secondary Outcome: Change in Three Domains of Men's Sexual Health Questionnaire (MSHQ)
Description: Men's Sexual Health Questionnaire (MSHQ), a 25-item questionnaire, assesses sexual function and satisfaction. It consists 5 domains: Erection (3 items, ranging from 0 to 15 (best)), Ejaculation (7 items, ranging from 1 to 35 (best)), Satisfaction (6 items, ranging from 6 to 30 (best)), Sexual desire (4 items, ranging 4-20 (best)), and Sexual activity (3 items, ranging 3-15 (best)). Erection, Ejaculation and Satisfaction domains were measured and the higher score representing better sexual function and satisfaction.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale
  Erection: number analyzed (Participants) | 30 | 20 | 34 | 10
  Erection | 0.80 (0.36) | 0.80 (0.52) | -0.65 (0.48) | 1.30 (0.45)
  Ejaculation: number analyzed (Participants) | 32 | 21 | 35 | 11
  Ejaculation | 1.34 (1.15) | 2.38 (1.72) | -1.46 (1.16) | -1.55 (3.26)
  Satisfaction: number analyzed (Participants) | 33 | 21 | 30 | 11
  Satisfaction | 1.03 (0.58) | 0.98 (0.85) | -0.40 (0.84) | 1.27 (1.05)

6. Secondary Outcome: Change in Two Domains of Expanded Prostate Cancer Index Composite (EPIC)
Description: Expanded Prostate Cancer Index Composite (EPIC) is a 50-item, comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Of its four domains, the sexual domain (range 0-100) and hormonal domain (range 0-100) were utilized. The response for each item is standardized to a 0 to 100 scale. Higher score yields better quality of life.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale
  Sexual function: number analyzed (Participants) | 32 | 24 | 34 | 12
  Sexual function | 1.86 (2.14) | 3.68 (3.04) | 0.08 (2.52) | 5.77 (3.90)
  Hormonal function: number analyzed (Participants) | 33 | 24 | 35 | 12
  Hormonal function | 1.24 (1.06) | 0.44 (2.04) | 0.52 (1.22) | 6.25 (5.79)

7. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale
Description: The FACIT Fatigue Scale is a 13-item questionnaire that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point scale (4 = not at all fatigued to 0 = very much fatigued). Score ranges 0-52. The higher the score, the better the quality of life.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale | 0.31 (1.30) | 2.29 (1.36) | -0.36 (1.28) | 0.26 (1.47)

8. Secondary Outcome: Change in Hypogonadism Energy Diary (HED)
Description: Hypogonadism Energy Diary (HED) is a 4-item questionnaire that intended to assess real-time energy levels. Score ranges 0 to100 with higher scores representing higher energy. each question uses an 11-point numerical rating scale (0-10) with 10 corresponding to full of energy or extreme tiredness. HED score was the average of the scores for these 4 items. Scores were linearly transformed to a 0 to 100 scale. Higher scores representing higher energy.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale | -0.45 (2.78) | 2.71 (2.82) | 2.64 (3.42) | 1.73 (5.07)

9. Secondary Outcome: Change in International Prostate Symptom Score (IPSS)
Description: International Prostate Symptom Score (IPSS) is a 8-item, extensively validated and widely used self-reported measure of lower urinary tract symptoms questionnaire. It includes Urinary Symptoms (item1-7, range 0-35) and Quality of Life Due to Urinary Symptoms (item 8, range 0-6). The higher the score, the severer of the urinary symptoms and worse quality of life due to symptoms.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale
  Urinary Symptoms | -0.30 (0.59) | -2.08 (0.65) | 0.06 (0.48) | 0.00 (0.62)
  Quality of Life Due to Urinary Symptoms: number analyzed (Participants) | 32 | 24 | 35 | 13
  Quality of Life Due to Urinary Symptoms | -0.13 (0.13) | -0.17 (0.17) | -0.03 (0.18) | -0.15 (0.19)

10. Secondary Outcome: Change in Positive and Negative Affect Scale (PANAS)
Description: The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (very slightly or not at all) to 5 (extremely). Score ranges 10-50 for both positive and negative affect. The higher scores represent higher levels of positive/negative affect.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
units on a scale
  Positive Affect | 0.91 (0.89) | 0.75 (1.84) | 1.42 (1.03) | -0.77 (0.89)
  Negative Affect | -1.70 (0.72) | -1.38 (0.58) | 0.42 (0.58) | -2.77 (1.49)

11. Secondary Outcome: Change in Body Mass Using DXA
Description: Whole body, appendicular, and trunk lean mass were measured using dual energy X- ray absorptiometry (DXA), calibrated using a soft tissue phantom before each scan.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 32 | 24 | 34 | 13
kg
  Appendicular Fat Mass | -0.06 (0.11) | -0.19 (0.10) | -0.36 (0.11) | -0.13 (0.11)
  Trunk Fat Mass | -0.00 (0.14) | -0.32 (0.18) | -0.38 (0.16) | -0.72 (0.19)
  Total Fat Mass | -0.05 (0.22) | -0.52 (0.24) | -0.75 (0.22) | -0.86 (0.27)
  Appendicular Lean Mass | -0.04 (0.10) | 0.15 (0.13) | 0.80 (0.13) | 1.05 (0.23)
  Trunk Lean Mass | 0.22 (0.12) | 0.20 (0.19) | 0.68 (0.19) | 0.88 (0.26)
  Total Lean Mass | 0.20 (0.16) | 0.33 (0.27) | 1.48 (0.28) | 1.92 (0.42)

12. Secondary Outcome: Change of Maximal Voluntary Muscle Strength
Description: The maximal voluntary muscle strength was measured in the leg press exercise using the 1-repetition method
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: N
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 17 | 10 | 18 | 7
N | -12.6 (55.0) | 108.1 (56.8) | 48.1 (29.4) | 103.5 (37.1)

13. Secondary Outcome: Change in Gait Speed in 6-minute Walk
Description: Tests of Physical Function and Task-Specific Performance measured by gait speed in 6-min walk
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: m/sec
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 28 | 20 | 31 | 10
m/sec | 0.05 (0.02) | 0.07 (0.02) | 0.08 (0.02) | 0.05 (0.03)

14. Secondary Outcome: Change of 50 Meters Walk Tests- Unloaded /Loaded
Description: Tests of Physical Function and Task-Specific Performance measured by 50-meter timed walk + 20% load carry. Physical Function was evaluated using test of 50-meter loaded walking speed. One test consisted of walking 50 meters as rapidly as possible without running (unloaded) while the second test required participants to carry a load equivalent to 20% of their baseline body weight evenly distributed in two canvas tote bags(loaded). Time was measured electronically with a digital clock. Speed in meters per second is calculated by the following: 50/time.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: m/sec
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 28 | 21 | 32 | 11
m/sec
  Unloaded: number analyzed (Participants) | 28 | 21 | 28 | 10
  Unloaded | 0.06 (0.03) | 0.12 (0.04) | 0.03 (0.02) | 0.07 (0.06)
  Loaded: number analyzed (Participants) | 21 | 16 | 20 | 9
  Loaded | 0.05 (0.03) | 0.13 (0.05) | 0.05 (0.04) | 0.09 (0.05)

15. Secondary Outcome: Change in Power of Stair Climbing Tests- Unloaded/Loaded
Description: Tests of Physical Function and Task-Specific Performance measured by Stair-climbing power +/- 20% load carry. Physical Function was evaluated using two tests of stair climb power using an indoor 12-step staircase. One test consisted of ascending the 12-steps as rapidly as possible without running (unloaded stair climb) while the second test required participants to carry a load equivalent to 20% of their baseline body weight evenly distributed in two canvas tote bags (loaded stair climb). Time to ascend the stairs was measured electronically with a digital clock and switch mats placed at the base of the steps and on the 12th step. Power in watts is calculated by the following: [body weight (kilograms) * distance (meters)/ (time/60)] /6.12.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: watts
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 28 | 21 | 32 | 11
watts
  Unloaded: number analyzed (Participants) | 24 | 15 | 22 | 7
  Unloaded | 12.8 (26.1) | 19.7 (19.6) | 1.8 (15.6) | 51.7 (21.9)
  Loaded: number analyzed (Participants) | 18 | 10 | 11 | 5
  Loaded | 0.22 (24.89) | -36.6 (24.9) | -9.8 (21.5) | 59.4 (42.3)

16. Secondary Outcome: Change in Serum Total Testosterone Level
Description: Serum total testosterone levels during screening was measured in the Quest Diagnostics Laboratory, Chantilly, VA, using liquid chromatography tandem mass spectrometry (LC-MS/MS) method certified by the Hormone Standardization Program for Testosterone (HoST) of the Centers for Disease Control and Prevention, Atlanta, Georgia.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
ng/dL | -6.5 (15.8) | -83.5 (21.3) | -172.3 (27.6) | -185.2 (46.0)

17. Secondary Outcome: Change in Free Testosterone Level
Description: Free testosterone level for screening was measured using an equilibrium dialysis method.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 32 | 22 | 35 | 13
pg/mL | 0.19 (0.15) | 0.59 (0.18) | 1.43 (0.20) | 1.62 (0.41)

18. Secondary Outcome: Change in Serum Sex Hormone-binding Globulin (SHBG) Level
Description: Serum SHBG level was measured using two-site directed immuno-chemiluminescence assays with sensitivity 2.5 nmol/L, and coefficients of variation less than 10% in low, medium and high range
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 30 | 21 | 35 | 13
nmol/L | 0.6 (1.0) | -9.6 (1.3) | -21.7 (2.1) | -24.2 (5.5)

19. Secondary Outcome: Change in Serum Luteinizing Hormone (LH) Level
Description: Serum LH level was measured using two-site directed immuno-chemiluminescence assays with sensitivity 0.1 U/L, and coefficients of variation less than 10% in low, medium and high range
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: mIU/mL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 32 | 22 | 35 | 13
mIU/mL | 0.23 (0.27) | 0.11 (0.23) | 0.72 (1.27) | -0.42 (0.47)

20. Secondary Outcome: Change in Estradiol Levels
Description: Estradiol level was measured by LC-MS/MS.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 32 | 22 | 35 | 13
pg/mL | -0.2 (1.5) | -1.1 (1.1) | -5.5 (1.1) | -7.9 (2.1)

21. Secondary Outcome: Change of White Blood Cell
Description: White Blood Cell was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: K/uL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
K/uL | -0.24 (0.15) | 0.30 (0.29) | -0.21 (0.19) | 0.32 (0.20)

22. Secondary Outcome: Change of Red Blood Cell
Description: Red Blood Cell was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: K/uL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
K/uL | -0.08 (0.04) | -0.05 (0.05) | 0.03 (0.03) | 0.06 (0.08)

23. Secondary Outcome: Change in Hematocrit
Description: Hematocrit was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: percentage of volume of red cells
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
percentage of volume of red cells | -0.61 (0.33) | -0.30 (0.51) | 0.44 (0.25) | 0.11 (0.89)

24. Secondary Outcome: Change in Hemoglobin
Description: Hemoglobin was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
g/dL | -0.32 (0.11) | -0.12 (0.16) | 0.09 (0.09) | -0.01 (0.25)

25. Secondary Outcome: Change of Mean Corpuscular Volume (MCV)
Description: Mean corpuscular volume was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: fL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
fL | 0.32 (0.30) | 0.44 (0.48) | 0.37 (0.31) | -1.08 (0.84)

26. Secondary Outcome: Change of Red Blood Cell Distribution Width (RDW)
Description: Red blood cell distribution width (RDW) was measured for safety monitoring. RDW was calculated with: standard deviation of the mean cell size divided by the mean corpuscular volume of the red cells multiplied by 100
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: percentage of variation of red cells
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
percentage of variation of red cells | 0.09 (0.14) | -0.15 (0.22) | 0.18 (0.10) | -0.44 (0.29)

27. Secondary Outcome: Change in Platelet Count
Description: Platelet count was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: K/uL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
K/uL | 0.67 (4.61) | 6.54 (5.13) | 13.5 (4.9) | 28.7 (4.1)

28. Secondary Outcome: Change of Aspartate Aminotransferase (AST)
Description: Aspartate aminotransferase was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
U/L | -1.24 (0.67) | -1.25 (0.81) | 2.33 (0.82) | 4.46 (2.03)

29. Secondary Outcome: Change of Alanine Aminotransferase (ALT)
Description: Alanine aminotransferase was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
U/L | -1.36 (0.89) | -3.46 (1.51) | 1.28 (1.37) | 5.46 (3.35)

30. Secondary Outcome: Change of Total Bilirubin
Description: Total Bilirubin was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
mg/dL | -0.13 (0.03) | -0.02 (0.03) | -0.16 (0.05) | -0.18 (0.04)

31. Secondary Outcome: Change in Serum Alkaline Phosphatase
Description: Serum alkaline phosphatase was measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
U/L | -2.94 (1.45) | -2.83 (1.55) | -8.97 (1.44) | -14.1 (3.2)

32. Secondary Outcome: Change of Lipid Panel
Description: Plasma lipids were measured for safety monitoring.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 35 | 13
mg/dL
  Total Cholesterol | -7.55 (2.53) | -15.1 (5.8) | -13.4 (4.5) | -14.9 (7.9)
  HDL | -2.55 (1.18) | -4.38 (1.21) | -12.6 (1.3) | -14.6 (3.0)
  LDL | -6.00 (2.10) | -7.13 (5.44) | 0.57 (4.05) | 3.92 (6.94)
  Triglycerides | 9.36 (8.66) | -23.5 (7.4) | -7.40 (4.57) | -31.7 (24.5)

33. Secondary Outcome: Change in Fasting Glucose Levels
Description: Glucose will be measured in a fasting serum sample at Quest Lab.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 33 | 24 | 36 | 13
mg/dL | 0.33 (1.74) | 0.04 (2.02) | -2.78 (1.44) | -8.54 (4.31)

34. Secondary Outcome: Change in Insulin
Description: Insulin will be measured using an immunoassay at Quest lab.
Time Frame: 12 weeks from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
Number analyzed (Participants) | 15 | 11 | 16 | 3
uIU/mL | -0.17 (0.93) | 0.36 (1.52) | -1.63 (0.68) | -1.00 (0.50)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | LY2452473 Dose 1 | LY2452473 Dose 2 | LY2452473 Dose 3
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/28 | 0/36 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/36 | 2/28 | 1/36 | 1/14
Other Adverse Events (participants affected / at risk) | 33/36 | 22/28 | 33/36 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | LY2452473 Dose 1 (N=28) | LY2452473 Dose 2 (N=36) | LY2452473 Dose 3 (N=14)
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Metastatic ocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal Cancer (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | LY2452473 Dose 1 (N=28) | LY2452473 Dose 2 (N=36) | LY2452473 Dose 3 (N=14)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 (4) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 | 0 | 0
Chest discomfort (Cardiac disorders) | 0 | 1 (2) | 0 | 0
Dizziness (Cardiac disorders) | 1 (3) | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Endocrine disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 2 (3) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 (5) | 1 | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Decreased appetite (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 1 | 2 | 1
Increased appetite (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 0
Night sweats (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Lyme Disease (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 2 (3) | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 | 1 | 3 (11)
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 (3) | 0 | 0
Hand injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Palate injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 (2)
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 (3) | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Biopsy skin (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Ankle impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 (3) | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 | 1 | 1
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 | 5 (8) | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 | 1 (2) | 0
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 (2) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (2) | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin laceration (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT02499497/Prot_SAP_000.pdf